CLINICAL TRIAL: NCT02966483
Title: Transanal Versus Laparoscopic Total Mesorectal Excision for Mid and Low Rectal Cancer (TaLaR): a Multicentre Randomised Clinical Trial
Brief Title: Transanal Versus Laparoscopic Total Mesorectal Excision for Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Peking Union Medical College Hospital (Other); The First Hospital of Jilin University (Other); RenJi Hospital (Other); Shengjing Hospital (Other); The Second People's Hospital of Yibin (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Nanchong Central Hospital (Other Government); Zunyi Medical College (Other); The First Affiliated Hospital of University of South China (Other); Xinqiao Hospital (Unknown); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Ruijin Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-RECTAl-2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Rectal Neoplasms Malignant; Surgery
Keywords: Rectal cancer; Laparoscopic surgery; Total mesorectal excision; Transanal; Multicentre randomised clinical trial
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Transanal or Laparoscopic Total Mesorectal Excision treat rectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transanal Total Mesorectal Excision (Experimental): The rectum is mobilized and resected transanally (from bottom to up) according to TME principles, via transanal platform (either rigid or flexible platform).An ideal TaTME is defined as the extraperitoneal portion of the rectum being mobilized from below.
  Interventions: Procedure: TaTME
- Laparoscopic Total Mesorectal Excision (Active Comparator): The traditional laparoscopic TME (LpTME) was performed via standard laparoscopic techniques, including multiple trocars and conventional laparoscopic instruments.
  Interventions: Procedure: LpTME

INTERVENTIONS:
Procedure: TaTME — Transanal Total Mesorectal Excision
  Other Names: Transanal TME
  Arms: Transanal Total Mesorectal Excision
Procedure: LpTME — Conventional Laparoscopic Total Mesorectal Excision
  Other Names: Laparoscopic TME
  Arms: Laparoscopic Total Mesorectal Excision

SUMMARY:
Laparoscopic surgery for rectal cancer has been successfully proven to be a non-inferior alternative regarding resection quality, and oncological outcomes of patients as compared to open surgery in mangy clinical trails. Moreover, laparoscopic surgery is advantageous over open surgery with regard to operative invasiveness, patient's recovery, and wound related complications. Thus, laparoscopic surgery has gained great popularity over the past decades. However, specifically for mid and low rectal cancer, laparoscopic surgery is technically demanding, which sometimes leads to high morbidity and unsatisfactory resection quality, especially in challenging cases such as bulky mesorectum, enlarged prostate, irradiated pelvis, etc. Under this circumstance, transanal total mesorectal excision (TaTME) , the so called "down-to-up" alternative, has emerged as a promising solution to these problems in recent years and more and more small studies have proven the feasibility and advantages of this technique, making it become a hot topic among both literature and conferences. However, TaTME is still at early birth, higher-level evidences, either multicentric, or comparative study with conventional surgery is strikingly lacking. Thus the investigators conduct this multicentre randomised clinical trial, comparing transanal TME versus laparoscopic TME for mid and low rectal cancer, aiming to prove the hypothesis that TaTME may achieve better resection quality and result in non-inferior oncological outcome, as well as short term operative morbidity and mortality.

DETAILED DESCRIPTION:
Background:In recent years, transanal mesorectal excision (TaTME) has emerged as a promising surgical alternative for rectal cancer, especially for mid and low rectal cancer. Theoretically, TaTME holds the potential advantage of providing better access to mobilize the distal rectum, and thus could achieve better pathologic outcomes, such as lower involved circumferential margin (CRM) and incomplete resected mesorectum, which could translate into better oncological outcome for the patients in the long term. However, until now, the feasibility and the non-inferiority (compared with laparoscopic total mesorectal excision, LpTME) of this technique has only been validated in studies with limitations of small sample size, retrospective nature.

Study Objective:This study aims to evaluate the TaTME technique compared with conventional laparoscopic rectal surgery, focusing on resection quality, as well as long-term survival results.

Study design This study is a prospective, multi-center, randomized, open-label, parallel group trial. The randomisation ratio of TaTME over LpTME will be 1:1. A central electronic data capture (EDC) system will be utilized for randomization, electronic CRF and data collection. All comparative analyses will be conducted on an "intention to treat" basis.

Sample size: Sample-size calculation of this trial based on 3-year DFS and 5-year OS; but the sample size according to 5-year OS was larger than that based on 3-year DFS. The expected 5-year OS among clinical stage I-III rectal cancer patients treated with laTME was 77·4%. Allowing a difference of 10% as the non-inferiority margin, 910 patients would be required to sufficiently declare taTME noninferior to laTME in 5-year OS based on a log-rank test with an α error of 2·5% (in a two-sided test) and power of 80%. Assuming a dropout rate of 20%, a total of 1114 patients were planned to enroll for this trial.

Study Endpoints:The primary end point of this study is 3-year disease-free survival (DFS) rate and a 5-year overall survival (OS) rate. Secondary endpoints include: 1) resection quality, mainly including circumferential involvement rate, and completeness of mesorectum. Resected specimen was pathologically processed and assessed at each center by trained and qualified pathologists independently.2)short term operative results such as morbidity and mortality, etc.; 3) long term oncological outcome such as local recurrence, and overall survival. Besides, functional outcome and quality of life are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

histologically proven rectal adenocarcinoma;

tumor located below the level of peritoneal reflection ;

diagnosis of rectal cancer amenable to curative surgery;

no evidence of distant metastases;

preoperative tumor stage within III;

no threaten mesorectal fascia (MRF)after neoadjuvant therapy;

no contraindication to laparoscopic surgery;

without history of other malignancies;

Written informed consent

Exclusion Criteria:

could not perform sphincter preservation surgery (requiring a Mile's procedure);

T4b tumor invading adjacent organs;

T1 tumors that can be locally resected

should take neoadjuvant therapy but refuse it;

recurrent cancer;

concurrent or previous diagnosis of invasive cancer within 5 years;

emergent surgery with intestinal obstruction or perforation;

history of colorectal surgery;

fecal incontinence;

history of inflammatory bowel disease;

with contraindications to general anaesthesia(ASA class 4 or 5);

pregnant or breast-feeding;

history of mental disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1114 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years
  Disease-free survival
Overall survival | 5 years
  Overall survival

SECONDARY OUTCOMES:
Positive circumferential resection margin (CRM) | 3 years
  Involved CRM (tumor cells <1mm)
Overall survival | 10 years
  Overall survival
Mesorectal completeness | 3 years
  The quality of the mesorectum or TME specimen (complete;nearly complete; incomplete)
Number of retrieved lymph nodes | 3 years
  Number of retrieved lymph nodes
Morbidity rate | 1 years
  Morbidity rate
Mortality rate | 1 years
  Mortality rate
Anorectal function outcomes | 3 years
  To evaluate defecating function with Wexner score
Sexual functional outcomes | 3 years
  To evaluate sexual function with IIEF(International Index of Erectile Function) questionnaire
The patient's Quality of life: EORTC QLQ-30 questionnaire | 3 years
  To evaluate quality of life with EORTC QLQ-30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wang, MD,PHD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (16):
- China (16):
  - Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Department of General Surgery, Daping Hospital, Army Medical university, Chongqing, Chongqing Municipality
  - Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Department of Gastrointestinal Surgery, The First Hospital of Jilin University, Changchun, Jilin
  - Department of Colorectal Surgery, Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Gastrointestinal Surgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University,, Shanghai, Shanghai Municipality
  - Department of Gastrointestinal Surgery，The Affiliated Nanchong Central Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Department of gastrointestinal surgery, the Second People's Hospital of Yibin, Yibin, Sichuan
  - XinQiao Hospital of Army Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen WH, Kang L, Luo SL, Zhang XW, Huang Y, Liu ZH, Wang JP. Transanal total mesorectal excision assisted by single-port laparoscopic surgery for low rectal cancer. Tech Coloproctol. 2015 Sep;19(9):527-34. doi: 10.1007/s10151-015-1342-1. Epub 2015 Jul 29. PMID 26220109
- [Background] Kang L, Chen WH, Luo SL, Luo YX, Liu ZH, Huang MJ, Wang JP. Transanal total mesorectal excision for rectal cancer: a preliminary report. Surg Endosc. 2016 Jun;30(6):2552-62. doi: 10.1007/s00464-015-4521-2. Epub 2015 Aug 27. PMID 26310534
- [Derived] Zeng Z, Luo S, Zhang H, Wu M, Ma D, Wang Q, Xie M, Xu Q, Ouyang J, Xiao Y, Song Y, Feng B, Xu Q, Wang Y, Zhang Y, Shi L, Ling L, Zhang X, Huang L, Yang Z, Peng J, Wu X, Ren D, Huang M, Lan P, Wang J, Tong W, Ren M, Liu H, Kang L; Chinese Transanal Endoscopic Surgery Collaborative (CTESC) Group. Transanal vs Laparoscopic Total Mesorectal Excision and 3-Year Disease-Free Survival in Rectal Cancer: The TaLaR Randomized Clinical Trial. JAMA. 2025 Mar 4;333(9):774-783. doi: 10.1001/jama.2024.24276. PMID 39847361
- [Derived] Chen M, Ye F, Huang P, Liang Z, Liu H, Zheng X, Li W, Luo S, Kang L, Huang L. Inflammatory stress response after transanal vs laparoscopic total mesorectal excision: a cohort study based on the TaLaR trial. Int J Surg. 2024 Jan 1;110(1):151-158. doi: 10.1097/JS9.0000000000000838. PMID 37916926
- [Derived] Zeng Z, Luo S, Chen J, Cai Y, Zhang X, Kang L. Comparison of pathological outcomes after transanal versus laparoscopic total mesorectal excision: a prospective study using data from randomized control trial. Surg Endosc. 2020 Sep;34(9):3956-3962. doi: 10.1007/s00464-019-07167-1. Epub 2019 Oct 4. PMID 31586244